CLINICAL TRIAL: NCT00570206
Title: An Evaluation of Motivational Interviewing to Increase Compliance in a Probation Setting (Enhancing Communication and Officer Responsivity; ENCORE)
Brief Title: An Evaluation of Motivational Interviewing to Increase Compliance in a Probation Setting
Acronym: ENCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Scott T. Walters, PhD, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SPH-07-0487; 07C71GJS8
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Compliance With Terms of Probation Sentence
Keywords: Probation; Motivational
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 1 (Experimental): Probation officers trained to use Motivational Interviewing while conducting meetings with probationers.
  Interventions: Behavioral: Motivational Interviewing
- 2 (No Intervention): Probation officers who are interested in Motivational Interviewing, but have not yet been trained to use it while conducting meetings with probationers.
- 3 (No Intervention): Treatment as usual. Regular probation officers conduct standard meetings with probationers.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Probation officers trained to use Motivational Interviewing while conducting meetings with probationers.
  Arms: 1

SUMMARY:
The purpose of this study is to examine the effects of Motivational Interviewing (MI) on probationer progress over a 6-month period, using probation officers as the MI providers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be on felony probation.
2. Participants must be English speaking.
3. Participants must be classified as medium or high-risk.
4. Participants must be placed on a non-specialized caseload.
5. Participants must be at least 18 years of age.

Exclusion Criteria:

1. Does not speak English.
2. Is less than 18 years old.
3. Is not on felony probation.
4. Is not classified as medium or high-risk.
5. Is placed on a specialized caseload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Revocations | 6 months
Absconder Status | 6 months
Urinalysis (UA) Data | 6 months
Arrest Data | 6 months

SECONDARY OUTCOMES:
Officer Responses Questionnaire | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Walters, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Dallas County Community Supervision and Corrections, Dallas, Texas
  - University of Texas School of Public Health Dallas Regional Campus, Dallas, Texas